CLINICAL TRIAL: NCT00150202
Title: Clinical Study Of EYE001 In Subfoveal Choroidal Neovascularization Secondary To Age-Related Macular Degeneration
Brief Title: Clinical Study Of EYE001 For Wet-Type AMD (Age-Related Macular Degeneration)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A5751010
Record Dates: First submitted 2005-09-06; First posted 2005-09-08 (Estimated); Last update posted 2007-05-07 (Estimated); Status verified 2006-11

CONDITIONS: Macular Degeneration
MeSH Terms: conditions — Macular Degeneration | interventions — pegaptanib

INTERVENTIONS:
Drug: pegaptanib sodium

SUMMARY:
This study will examine the efficacy and safety of pegaptanib sodium in Japanese patients with wet-type AMD, in order to establish that there is no large difference in the efficacy and the safety of the drug between Western and Japanese patients.

ELIGIBILITY:
Inclusion Criteria:

* Wet AMD, Visual Acuity from 20/320 to 20/40

Exclusion Criteria:

* Diabetic retinopathy, laser coagulation history

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90
Dates: Start 2004-07; Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
Visual aquity change from the baseline to 54 weeks after the first treatment is expected to be similar to that seen in the Western studies.

SECONDARY OUTCOMES:
Safety profile of pegaptanib including side effects and lab test from the baseline to 54 weeks after the first treatment. Blood concentration of the drug from the baseline to 54 weeks after the irst treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (14):
- Japan (14):
  - Pfizer Investigational Site, Nagoya, Aichi-ken
  - Pfizer Investigational Site, Urayasu-shi, Chiba
  - Pfizer Investigational Site, Tokyo, Chiyoda-ku
  - Pfizer Investigational Site, Fukuoka, Fukuoka
  - Pfizer Investigational Site, Fukushima, Fukushima
  - Pfizer Investigational Site, Maebashi, Gunma
  - Pfizer Investigational Site, Sapporo, Hokkaido
  - Pfizer Investigational Site, Kida-gun, Kagawa-ken
  - Pfizer Investigational Site, Kyoto, Kyoto
  - Pfizer Investigational Site, Moriguchi, Osaka
  - Pfizer Investigational Site, Suita, Osaka
  - Pfizer Investigational Site, Ōtsu, Shiga
  - Pfizer Investigational Site, Mitaka, Tokyo
  - Pfizer Investigational Site, Shinjuku-ku, Tokyo